CLINICAL TRIAL: NCT06759532
Title: Prognostic Role of Persistent Microvascular Obstruction by Cardiac Magnetic Resonance for ST-segment Elevation Myocardial Infarction
Brief Title: Impact of Persistent Microvascular Obstruction by Cardiac Magnetic Resonance on Prognosis for ST-segment Elevation Myocardial Infarction
Acronym: IMCOME
Status: Completed | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Qian geng, MD, Chinese PLA General Hospital
Other Study IDs: Persistent MVO on prognosis; Z-2017-26-2202-2 (Other Grant/Funding Number: China international medical fundation)
Record Dates: First submitted 2024-12-30; First posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-12

CONDITIONS: ST Elevation (STEMI) Myocardial Infarction
Keywords: Microvascular occlusion;; ST-segment elevation myocardial infarction; Prognosis
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Without MVO group: STEMI patients without MVO both in the acutephase and chronic phase of myocardial inarction
- with transient MVO group: STEMI patients with MVO only in the acutephase of myocardial inarction
- with persietent MVO group: STEMI patients without MVO both in the acutephase and chronic phase of myocardial inarction

SUMMARY:
The aims of the study were to evaluate the predictive value of persistent microvascular obstruction (MVO) by cardiac magnetic resonance for main adverse cardiac events in ST-segment elevation myocardial infarction patients.

MVO in the acute phase of myocardial infarction has been considered to be strong predictor of a poor prognosis. We plan to explore the relationship between persistent MVO and the long-term prognosis of patients with STEMI. We made hypothesis that patients with persistent MVO have a poor prognosis.

ELIGIBILITY:
Inclusion Criteria:

* ST-segment elevation myocardial infarction undewent primary percutaneous coronary intervention

Exclusion Criteria:

* contraindications for cardiac magnetic resonance
* severe heart failure
* previous myocardial infarction.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients in this study were diagnosis as STEMI, and were plan to undergo primary percutaneous coronary intervention and were plan to underwent cardiac magnetic resonance at 7 days and 6 months after primary percutaneous coronary intervention . The patients were divided into three groups according to the presence of absence of MVO at the first cardiac magnetic resonance and second cardiac magnetic resonance.
Sampling Method: Probability Sample
Enrollment: 344 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2024-07-20 (Actual); Study Completion 2024-10-20 (Actual)

PRIMARY OUTCOMES:
Main aderverse cardiac events | 5 years after myocardiac infarction
  Composite endpoint of all-cause death, readmission due to heart failure, recurrent myocardial infarction, and unexpected vascularization.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA general hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Symons R, Pontone G, Schwitter J, Francone M, Iglesias JF, Barison A, Zalewski J, de Luca L, Degrauwe S, Claus P, Guglielmo M, Nessler J, Carbone I, Ferro G, Durak M, Magistrelli P, Lo Presti A, Aquaro GD, Eeckhout E, Roguelov C, Andreini D, Vogt P, Guaricci AI, Mushtaq S, Lorenzoni V, Muller O, Desmet W, Agati L, Janssens S, Bogaert J, Masci PG. Long-Term Incremental Prognostic Value of Cardiovascular Magnetic Resonance After ST-Segment Elevation Myocardial Infarction: A Study of the Collaborative Registry on CMR in STEMI. JACC Cardiovasc Imaging. 2018 Jun;11(6):813-825. doi: 10.1016/j.jcmg.2017.05.023. Epub 2017 Aug 16. PMID 28823746
- [Background] Bodi V, Gavara J, Lopez-Lereu MP, Monmeneu JV, de Dios E, Perez-Sole N, Bonanad C, Marcos-Garces V, Canoves J, Minana G, Nunez J, Moratal D, Chorro FJ, Rodriguez-Palomares JF, Freixa A, Borras R, Ortiz-Perez JT, Rios-Navarro C. Impact of Persistent Microvascular Obstruction Late After STEMI on Adverse LV Remodeling: A CMR Study. JACC Cardiovasc Imaging. 2023 Jul;16(7):919-930. doi: 10.1016/j.jcmg.2023.01.021. Epub 2023 Apr 12. PMID 37052556
- [Background] Lechner I, Reindl M, Stiermaier T, Tiller C, Holzknecht M, Oberhollenzer F, von der Emde S, Mayr A, Feistritzer HJ, Carberry J, Carrick D, Bauer A, Thiele H, Berry C, Eitel I, Metzler B, Reinstadler SJ. Clinical Outcomes Associated With Various Microvascular Injury Patterns Identified by CMR After STEMI. J Am Coll Cardiol. 2024 May 28;83(21):2052-2062. doi: 10.1016/j.jacc.2024.03.408. PMID 38777509
- [Background] Orn S, Manhenke C, Greve OJ, Larsen AI, Bonarjee VV, Edvardsen T, Dickstein K. Microvascular obstruction is a major determinant of infarct healing and subsequent left ventricular remodelling following primary percutaneous coronary intervention. Eur Heart J. 2009 Aug;30(16):1978-85. doi: 10.1093/eurheartj/ehp219. Epub 2009 Jun 6. PMID 19502624
- [Background] Bodi V, Sanchis J, Lopez-Lereu MP, Nunez J, Sanz R, Palau P, Gomez C, Moratal D, Chorro FJ, Llacer A. Microvascular perfusion 1 week and 6 months after myocardial infarction by first-pass perfusion cardiovascular magnetic resonance imaging. Heart. 2006 Dec;92(12):1801-7. doi: 10.1136/hrt.2005.077305. Epub 2006 Jun 27. PMID 16803939
- [Background] Weir RA, Murphy CA, Petrie CJ, Martin TN, Balmain S, Clements S, Steedman T, Wagner GS, Dargie HJ, McMurray JJ. Microvascular obstruction remains a portent of adverse remodeling in optimally treated patients with left ventricular systolic dysfunction after acute myocardial infarction. Circ Cardiovasc Imaging. 2010 Jul;3(4):360-7. doi: 10.1161/CIRCIMAGING.109.897439. Epub 2010 Mar 26. PMID 20348438
- [Background] van Kranenburg M, Magro M, Thiele H, de Waha S, Eitel I, Cochet A, Cottin Y, Atar D, Buser P, Wu E, Lee D, Bodi V, Klug G, Metzler B, Delewi R, Bernhardt P, Rottbauer W, Boersma E, Zijlstra F, van Geuns RJ. Prognostic value of microvascular obstruction and infarct size, as measured by CMR in STEMI patients. JACC Cardiovasc Imaging. 2014 Sep;7(9):930-9. doi: 10.1016/j.jcmg.2014.05.010. PMID 25212799
- [Background] Rios-Navarro C, Marcos-Garces V, Bayes-Genis A, Husser O, Nunez J, Bodi V. Microvascular Obstruction in ST-Segment Elevation Myocardial Infarction: Looking Back to Move Forward. Focus on CMR. J Clin Med. 2019 Oct 28;8(11):1805. doi: 10.3390/jcm8111805. PMID 31661823